CLINICAL TRIAL: NCT05073679
Title: A Double-Blind Placebo-Controlled Evaluation of Effectiveness of Oral Naltrexone in Management of Adolescent Eating Disorders
Brief Title: Oral Naltrexone In Pediatric Eating Disorders
Acronym: ONPED
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low enrollment numbers, pharmacy not able to acquire sufficient study article component (methylcellulose) due to manufacturer backorder
Sponsor: Rosemary Claire Roden (Other)
Collaborators: Children's Miracle Network (Other)
Responsible Party: Sponsor-Investigator, Rosemary Claire Roden, Assistant Professor of Pediatrics, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00014382; 150408 (Other: Food and Drug Administration)
Record Dates: First submitted 2021-07-19; First posted 2021-10-11 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Anorexia Nervosa/Bulimia; Anorexia in Adolescence; Anorexia Nervosa, Atypical; Anorexia Nervosa, Binge Eating/Purging Type; Purging (Eating Disorders); Impulsive Behavior; Eating Disorders; Bulimia Nervosa; Eating Disorders in Adolescence
MeSH Terms: conditions — Anorexia Nervosa; Bulimia; Feeding and Eating Disorders; Impulsive Behavior; Bulimia Nervosa | interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: double-blind, placebo controlled randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Penn State Health IDS pharmacy will purchase Naltrexone 50mg tablets from a pharmaceutical wholesaler. The IDS pharmacy will purchase gelatin capsules and USP grade methylcellulose from a pharmacy supplier to be used for compounding the active and placebo capsules. For the active Naltrexone 50mg capsules, a Naltrexone 50mg tablet will be placed in an empty gelatin capsule with methylcellulose filler. The placebo capsules will be empty gelatin capsules filled with Methylcellulose.
  Participants will be randomized using redcap at enrollment to either study article or placebo, and neither investigators nor care providers will be aware of which article the participants receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Oral naltrexone, to start as 25mg for three days then 50mg a day for 6 weeks. Oral naltrexone generic tabs will be blinded in opaque gelatin capsules with methylcellulose filler
  Interventions: Drug: Naltrexone Hydrochloride
- Control (Placebo Comparator): Opaque gelatin capsules with methylcellulose filler, taken by mouth once a day for six weeks
  Interventions: Other: Control

INTERVENTIONS:
Drug: Naltrexone Hydrochloride — 25mg x 3 days then 50mg a day thereafter
  Arms: Intervention
Other: Control — Methylcellulose and gelatin capsule only
  Arms: Control

SUMMARY:
The objective of this study is to evaluate the effectiveness of oral naltrexone tablets in pediatric and adolescent eating disorders, in particular anorexia nervosa and bulimia nervosa, as compared to placebo. Study participants will be patients in a partial hospitalization program or intensive outpatient program for eating disorder.

DETAILED DESCRIPTION:
Subjects participating in this study will receive routine care for eating disorder at a partial hospitalization (PHP) level of care at MSHMC. In PHP, all patients have weekly medical screening visits for the duration of their time in care, as well as weekly individual therapy sessions, individual dietician sessions, and psychiatry appointments. They have supervised meals and numerous group therapy sessions. Every three weeks, patients in PHP complete a battery of mood and eating disorder indices including those evaluated in this study; participants in this study will complete an additional two surveys with this routine battery. Participants in this study will have no alterations in their routine eating disorder care outside of study article use and these additional surveys.

Subjects will be enrolled at their first visit for eating disorder programming at child or adult partial hospitalization (PHP) programming at MSHMC adolescent medicine eating disorders clinic. Informed consent/assent will be obtained as described above.

The subject will be provided with oral naltrexone or placebo weekly from the MSHMC research pharmacy. Subjects will be given one weeks' worth of medication at a time. Subjects will be randomized at enrollment to receive either study drug (naltrexone) or placebo. Participants or parents of minor participants will be provided study drug or placebo following completion of urine drug screen and consent/assent. Patients will take the medication daily for six weeks. For subjects who are enrolled in child PHP and who eat meals with parents, the families may choose to administer study drug during meals at programming. For adult patients enrolled in adult programming, subjects may choose to self-administer the medication.

On their first contact with PHP, all patients in Child PHP complete various eating disorder indices as a part of routine care, including the ED-15, EDE-Q, RCMAS, CDI, GAD-7, and PHQ-9. This battery of indices is repeated every 3 weeks while a patient is in programming.

For those who are enrolled in this study, they will complete their routine indices, in addition they will also complete the BIS/BAS and the ABUSI at enrollment and at weeks 3, 6, and 9 (after completion of medication) while in programming. Participants will receive routine eating disorder care while in PHP.

Patients in Adult PHP typically complete a different inventory every three weeks. If a patient chooses to participate in this study they will be asked to complete the same surveys as participants in Child PHP, and they will receive the same amount and type of compensation.

Six months after enrollment, subjects will be sent copies of ED-15, EDE-Q, GAD-7, PHQ-9, BIS/BAS, and ABUSI indices either in an in-person medical appointment or via RedCap to complete. If the patient returns for medical follow-up between 5 and 7 months after enrollment, their height, weight, and body mass index will also be recorded to determine if weight restoration was maintained.

At initial contact with the eating disorders clinic, all patients receive an initial battery of laboratory tests as a part of the standard of care for eating disorder. These tests include liver function assays and transaminase levels.

ELIGIBILITY:
Inclusion Criteria:

* Ages 13-25 (inclusive)
* Any sex
* Diagnoses of anorexia nervosa binge-purge subtype, bulimia nervosa, purging disorder, or atypical anorexia nervosa with bingeing or purging behaviors according to the Diagnostic and Statistical Manual version 5 diagnostic criteria
* Electing to participate in child or adult partial hospitalization program for eating disorder treatment at MSHMC

The diagnostic criteria for anorexia nervosa, binge-purge subtype, are:

A. Restriction of energy intake relative to requirements, leading to a significantly low body weight in the context of age, sex, developmental trajectory, and physical health. Significantly low weight is defined as a weight that is less than minimally normal or, for children and adolescents, less than minimally expected.

B. Intense fear of gaining weight or of becoming fat, or persistent behavior that interferes with weight gain, even though at a significantly low weight.

C. Disturbance in the way in which one's body weight or shape is experienced, undue influence of body weight or shape on self-evaluation, or persistent lack of recognition of the seriousness of the current low body weight D. During the last three months the individual has engaged in recurrent episodes of binge eating or purging behaviour (i.e. self-induced vomiting, or the misuse of laxatives, diuretics, or enemas).19 E. A diagnosis of atypical anorexia nervosa can be made when the body weight is normal or high If these patients engage in bingeing or purging behaviors as defined in anorexia nervosa, binge-purge subtype, they are eligible for inclusion in this study

The diagnostic criteria for bulimia nervosa are:

A. Recurrent episodes of binge eating. An episode of binge eating is characterized by

B. both:

i. Eating in a discrete period of time (e.g. within any 2 hour period), an amount of food that is definitely larger than what most individuals would eat in a similar period of time under similar circumstances; ii. A sense of lack of control over eating during the episodes (e.g. a feeling that one cannot stop eating or control what or how much one is eating.

C. Recurrent inappropriate compensatory behaviors to prevent weight gain, such as self-induced vomiting; misuse of laxatives, diuretics, or other medications; fasting; or excessive exercise.

D. The binge eating and inappropriate compensatory behaviors both occur, on average, at least once a week for 3 months.

E. Self-evaluation is unduly influenced by body shape and weight. F. The disturbance does not occur exclusively during episodes of anorexia nervosa.

• The diagnostic criteria for purging disorder are: recurrent purging behavior to influence weight or shape (e.g. self-induced vomiting; misuse of laxatives, diuretics, or other medications) in the absence of binge eating.

Exclusion Criteria:

* Diagnosis of intellectual disability
* History of known genetic or neurologic disease
* Need for treatment with opioid painkillers
* Weight <25kg
* Inability to swallow pills
* Lack of proficiency in written or spoken English
* Urine drug screen positive for opioids at enrollment
* Positive serum pregnancy test at enrollment
* Lactation
* Elevation of three times the upper limit of normal for age in either alanine aminotransferase (ALT) or asparagine aminotransferase (AST).High risk of suicide at enrollment on Columbia Suicide Severity Rating Scale (C-SSRS, for participants age 18-25) or Ask Suicide Screening Questions (ASQ, participants age 13 to 17)

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary C Roden, MD, Principal Investigator — PennState Health Children's Hospital
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No participant data is planned to be shared at the moment to protect patient privacy, as participants are all enrolled in a partial hospitalization program for mental health conditions.

REFERENCES:
- [Background] Tatham M, Turner H, Mountford VA, Tritt A, Dyas R, Waller G. Development, psychometric properties and preliminary clinical validation of a brief, session-by-session measure of eating disorder cognitions and behaviors: The ED-15. Int J Eat Disord. 2015 Nov;48(7):1005-15. doi: 10.1002/eat.22430. Epub 2015 May 26. PMID 26011054
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Smucker MR, Craighead WE, Craighead LW, Green BJ. Normative and reliability data for the Children's Depression Inventory. J Abnorm Child Psychol. 1986 Mar;14(1):25-39. doi: 10.1007/BF00917219. PMID 3950219
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Horowitz LM, Bridge JA, Teach SJ, Ballard E, Klima J, Rosenstein DL, Wharff EA, Ginnis K, Cannon E, Joshi P, Pao M. Ask Suicide-Screening Questions (ASQ): a brief instrument for the pediatric emergency department. Arch Pediatr Adolesc Med. 2012 Dec;166(12):1170-6. doi: 10.1001/archpediatrics.2012.1276. PMID 23027429
- [Background] Campbell K, Peebles R. Eating disorders in children and adolescents: state of the art review. Pediatrics. 2014 Sep;134(3):582-92. doi: 10.1542/peds.2014-0194. PMID 25157017
- [Derived] Roden RC, Billman M, Lane-Loney S, Essayli J, Mahr F, Vrana K, Ryan S. An experimental protocol for a double-blind placebo-controlled evaluation of the effectiveness of oral naltrexone in management of adolescent eating disorders. Contemp Clin Trials. 2022 Nov;122:106937. doi: 10.1016/j.cct.2022.106937. Epub 2022 Sep 24. PMID 36167287
- See also: Oral naltrexone package insert — https://www.accessdata.fda.gov/drugsatfda_docs/label/2013/018932s017lbl.pdf
- See also: DSM-5 Chapter on Feeding and Eating Disorders — https://www.researchgate.net/publication/258253416_Feeding_and_Eating_Disorders_in_DSM-5

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 16 [14 to 17] | 17 [15.25 to 19.25] | 16.5 [14 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 1 | 5
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic | 5 | 1 | 6
  Hispanic | 0 | 0 | 0
  Multiple | 0 | 1 | 1
  Unknown | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: ED-15 Score
Description: ED-15 is an evidenced-based metric of eating disorder symptom severity and frequency. The global score ranges from a 0 to 6 with higher scores indicating more eating disordered psychopathology.
Time Frame: Time Frame: Measured at the following timepoints: enrollment
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 3.5 (2.016184515) | 4.7 (0.871779789)

2. Primary Outcome: ED-15 Score
Description: as for outcome 1
Time Frame: Time Frame: Measured at the following timepoints: one week
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 3.08 (1.845806057) | 4.675 (0.784750491)

3. Primary Outcome: ED-15 Score
Description: as for outcome 1
Time Frame: Time Frame: Measured at the following timepoints: three week
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 3.04 (1.820164828) | 4.025 (1.508586535)

4. Primary Outcome: ED-15 Score
Description: as for outcome 1
Time Frame: Time Frame: Measured at the following timepoints: six weeks
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 3
score on a scale | 1.825 (1.701714821) | 3.5 (2.364318084)

5. Primary Outcome: ED-15 Score
Description: as for outcome 1
Time Frame: Time Frame: Measured at the following timepoints: nine weeks (last week of treatment)
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 1
score on a scale | 1.075 (0.736545993) | 4.5 (0)

6. Primary Outcome: ED-15 Score
Description: as for outcome 1
Time Frame: Time Frame: Measured at the following timepoints: 6 months after enrollment
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 1
score on a scale | 0.866666667 (0.776745347) | 4.3 (0)

7. Secondary Outcome: Eating Disorder Examination Questionnaire Score (EDE-Q)
Description: EDE-Q is an evidence-based metric of eating disorder severity. The global EDE-Q score ranges from 0 to 6, with higher scores indicating a higher eating disorder psychopathology.
Time Frame: Measured at the following timepoints: enrollment
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 3.3925 (1.8216) | 4.72031 (0.806764613)

8. Secondary Outcome: Eating Disorder Examination Questionnaire Score (EDE-Q)
Description: as for outcome 7
Time Frame: Measured at the following timepoints: one week
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 2.87 (1.744810385) | 4.315625 (0.645285386)

9. Secondary Outcome: Eating Disorder Examination Questionnaire Score (EDE-Q)
Description: as for outcome 7
Time Frame: Measured at the following timepoints: three weeks
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 2.66375 (1.553369573) | 3.9953125 (1.634008483)

10. Secondary Outcome: Eating Disorder Examination Questionnaire Score (EDE-Q)
Description: as for outcome 7
Time Frame: Measured at the following timepoints: six weeks
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 3
score on a scale | 1.6546875 (1.524132053) | 3.2 (2.385773263)

11. Secondary Outcome: Eating Disorder Examination Questionnaire Score (EDE-Q)
Description: as for outcome 7
Time Frame: Measured at the following timepoints: nine weeks (last week of treatment)
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 1
score on a scale | 0.753125 (0.538770301) | 4.04375 (0)

12. Secondary Outcome: Eating Disorder Examination Questionnaire Score (EDE-Q)
Description: as for outcome 7
Time Frame: Measured at the following timepoints: 6 months after enrollment
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 1
score on a scale | 2.4125 (0.724577822) | 3.90625 (0)

13. Secondary Outcome: Patient Health Questionnaire Score (PHQ-9)
Description: Evidence-based metric of depression, min = 0, max= 27, higher scores indicate more severe depression
Time Frame: Measured at the following timepoints: enrollment
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 13.8 (8.043631021) | 12 (4.966554809)

14. Secondary Outcome: Patient Health Questionnaire Score (PHQ-9)
Description: Evidence-based metric of depression, min = 0, max= 27, higher scores indicate more severe depression
Time Frame: Measured at the following timepoints: one week
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 12.8 (8.167006796) | 11.5 (4.203173404)

15. Secondary Outcome: Patient Health Questionnaire Score (PHQ-9)
Description: Evidence-based metric of depression, min = 0, max= 27, higher scores indicate more severe depression
Time Frame: Measured at the following timepoints: three weeks
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 10.4 (6.268971207) | 10.75 (4.991659711)

16. Secondary Outcome: Patient Health Questionnaire Score (PHQ-9)
Description: Evidence-based metric of depression, min = 0, max= 27, higher scores indicate more severe depression
Time Frame: Measured at the following timepoints: six weeks
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 3
score on a scale | 7.5 (4.434711565) | 10.66666667 (2.309401077)

17. Secondary Outcome: Patient Health Questionnaire Score (PHQ-9)
Description: Evidence-based metric of depression, min = 0, max= 27, higher scores indicate more severe depression
Time Frame: Measured at the following timepoints: nine weeks (last week of treatment)
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 2
score on a scale | 5.5 (6.191391874) | 12.5 (9.192388155)

18. Secondary Outcome: Patient Health Questionnaire Score (PHQ-9)
Description: Evidence-based metric of depression, min = 0, max= 27, higher scores indicate more severe depression
Time Frame: Measured at the following timepoints: 6 months after enrollment
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 1
score on a scale | 4.666666667 (5.507570547) | 4 (0)

19. Secondary Outcome: Generalized Anxiety Disorder Screener Score (GAD-7)
Description: evidence-based metric of anxiety, min=0, max=21, higher scores indicate more severe anxiety
Time Frame: Measured at the following timepoints: enrollment
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 10.8 (3.271085447) | 13.75 (5.560275773)

20. Secondary Outcome: Generalized Anxiety Disorder Screener Score (GAD-7)
Description: evidence-based metric of anxiety, min=0, max=21, higher scores indicate more severe anxiety
Time Frame: Measured at the following timepoints: one week
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 7.4 (3.577708764) | 12.75 (4.716990566)

21. Secondary Outcome: Generalized Anxiety Disorder Screener Score (GAD-7)
Description: evidence-based metric of anxiety, min=0, max=21, higher scores indicate more severe anxiety
Time Frame: Measured at the following timepoints: three weeks
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 6.8 (4.438468204) | 11 (4.69041576)

22. Secondary Outcome: Generalized Anxiety Disorder Screener Score (GAD-7)
Description: evidence-based metric of anxiety, min=0, max=21, higher scores indicate more severe anxiety
Time Frame: Measured at the following timepoints: six weeks
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 3
score on a scale | 6.75 (4.645786622) | 10.33333333 (3.511884584)

23. Secondary Outcome: Generalized Anxiety Disorder Screener Score (GAD-7)
Description: evidence-based metric of anxiety, min=0, max=21, higher scores indicate more severe anxiety
Time Frame: Measured at the following timepoints: nine weeks (last week of treatment)
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 2
score on a scale | 6 (6.976149845) | 9 (5.656854249)

24. Secondary Outcome: Generalized Anxiety Disorder Screener Score (GAD-7)
Description: evidence-based metric of anxiety, min=0, max=21, higher scores indicate more severe anxiety
Time Frame: Measured at the following timepoints: 6 months after enrollment
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 1
score on a scale | 5.666666667 (1.154700538) | 6 (0)

25. Secondary Outcome: Alexian Brothers Urge to Self-Injure Scale (ABUSI)
Description: evidence-based metric of urge to self-harm. min = 0 max = 30. Higher scores represent more intense urges to self-injure
Time Frame: Measured at the following timepoints: enrollment
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 3.4 (3.435112807) | 7.25 (7.632168761)

26. Secondary Outcome: Alexian Brothers Urge to Self-Injure Scale (ABUSI)
Description: evidence-based metric of urge to self-harm. min = 0 max = 30. Higher scores represent more intense urges to self-injure
Time Frame: Measured at the following timepoints: one week
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 3.6 (4.098780306) | 5.75 (4.924428901)

27. Secondary Outcome: Alexian Brothers Urge to Self-Injure Scale (ABUSI)
Description: evidence-based metric of urge to self-harm. min = 0 max = 30. Higher scores represent more intense urges to self-injure
Time Frame: Measured at the following timepoints: three weeks
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 2.8 (2.387467277) | 4.5 (3.415650255)

28. Secondary Outcome: Alexian Brothers Urge to Self-Injure Scale (ABUSI)
Description: evidence-based metric of urge to self-harm. min = 0 max = 30. Higher scores represent more intense urges to self-injure
Time Frame: Measured at the following timepoints: six weeks
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 3
score on a scale | 2.25 (2.62995564) | 11 (6.08276253)

29. Secondary Outcome: Alexian Brothers Urge to Self-Injure Scale (ABUSI)
Description: evidence-based metric of urge to self-harm. min = 0 max = 30. Higher scores represent more intense urges to self-injure
Time Frame: Measured at the following timepoints: nine weeks (last week of treatment)
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 2
score on a scale | 1.5 (3) | 9 (12.72792206)

30. Secondary Outcome: Alexian Brothers Urge to Self-Injure Scale (ABUSI)
Description: evidence-based metric of urge to self-harm. min = 0 max = 30. Higher scores represent more intense urges to self-injure
Time Frame: Measured at the following timepoints: 6 months after enrollment
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 1
score on a scale | 0.333333333 (0.577350269) | 0 (0)

31. Secondary Outcome: Barratt Impulsiveness Scale (BIS-11)
Description: Evidence-based metric of impulsivity. min = 30 max = 120. higher scores indicate higher levels of impulsivity.
Time Frame: Measured at the following timepoints: enrollment
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 62.2 (14.44645285) | 72.25 (9.569918147)

32. Secondary Outcome: Barratt Impulsiveness Scale (BIS-11)
Description: Evidence-based metric of impulsivity. min = 30 max = 120. higher scores indicate higher levels of impulsivity.
Time Frame: Measured at the following timepoints: one week
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 64 (17.88854382) | 71 (6.976149845)

33. Secondary Outcome: Barratt Impulsiveness Scale (BIS-11)
Description: Evidence-based metric of impulsivity. min = 30 max = 120. higher scores indicate higher levels of impulsivity.
Time Frame: Measured at the following timepoints: three weeks
Population: Numbers represent participants enrolled at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 4
score on a scale | 64.4 (12.77888884) | 69.5 (5.744562647)

34. Secondary Outcome: Barratt Impulsiveness Scale (BIS-11)
Description: Evidence-based metric of impulsivity. min = 30 max = 120. higher scores indicate higher levels of impulsivity.
Time Frame: Measured at the following timepoints: six weeks
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 3
score on a scale | 65.25 (14.22146265) | 69.66666667 (6.506407099)

35. Secondary Outcome: Barratt Impulsiveness Scale (BIS-11)
Description: Evidence-based metric of impulsivity. min = 30 max = 120. higher scores indicate higher levels of impulsivity.
Time Frame: Measured at the following timepoints: nine weeks (last week of treatment)
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 2
score on a scale | 63.25 (14.97497913) | 71 (12.72792206)

36. Secondary Outcome: Barratt Impulsiveness Scale (BIS-11)
Description: Evidence-based metric of impulsivity. min = 30 max = 120. higher scores indicate higher levels of impulsivity.
Time Frame: Measured at the following timepoints: 6 months after enrollment
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 1
score on a scale | 64 (10.58300524) | 60 (0)

37. Secondary Outcome: Percent of Weight Restoration
Description: For participants who need to restore weight, will evaluate the percent of weight gain in care
Time Frame: Will evaluate total percent of weight restoration via chart review at 9 weeks
Population: Numbers reflect participants enrolled at this time point. Other participants are lost to follow-up.
Measure: Mean (Standard Deviation); unit: percentage of weight restoration
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 2
percentage of weight restoration | 100.25 (5.068) | 94 (12)

38. Secondary Outcome: Percent of Weight Restoration
Description: For participants who need to restore weight, will evaluate the percent of weight gain in care
Time Frame: Will evaluate total percent of weight restoration via chart review 6 months after enrollment at about 33 weeks
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: percentage of weight restoration
Arm/Group | Intervention | Control
Number analyzed (Participants) | 2 | 2
percentage of weight restoration | 100.5 (10.60660172) | 84.5 (7.778174593)

39. Secondary Outcome: Need For Higher Level of Care
Description: Need to leave the current level of care (where the study is being conducted) to go to a residential, inpatient, or hospital facility
Time Frame: Will evaluate need for higher level of care at nine weeks
Population: We collected data for 8 out of 9 participants because an in-person visit was required for this variable to be evaluated. One participant was lost to follow-up and did not have an in-person visit at this time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 4
Participants
  Need for Higher Level of Care | 0 | 0
  No Need for Higher Level of Care | 4 | 4

40. Secondary Outcome: Need For Higher Level of Care
Description: as for outcome 39
Time Frame: Will evaluate need for higher level of care at 6 months after the end of the study at about 33 weeks
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 2 | 1
Participants
  Need for Higher Level of Care | 0 | 1
  No Need for Higher Level of Care | 2 | 0

41. Other Pre Specified Outcome: Columbia Suicide Severity Rating Scale (CSSRS)
Description: Evidence-based metric evaluating for presence of suicidal ideation and severity. Scores range from 1 (low risk) to 3 (high risk).
Time Frame: Measured at enrollment for patients age 17 or older
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1 | 2
Participants
  Low Risk | 0 | 1
  Medium Risk | 1 | 1
  High Risk | 0 | 0

42. Other Pre Specified Outcome: Columbia Suicide Severity Rating Scale (CSSRS)
Description: as for outcome 41
Time Frame: week 1 for patients age 17 or older
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1 | 2
Participants
  Low Risk | 1 | 1
  Medium Risk | 0 | 1
  High Risk | 0 | 0

43. Other Pre Specified Outcome: Columbia Suicide Severity Rating Scale (CSSRS)
Description: as for outcome 41
Time Frame: week 2 for patients age 17 or older
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1 | 2
Participants
  Low Risk | 0 | 1
  Medium Risk | 1 | 1
  High Risk | 0 | 0

44. Other Pre Specified Outcome: Columbia Suicide Severity Rating Scale (CSSRS)
Description: as for outcome 41
Time Frame: week 3 for patients age 17 or older
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1 | 2
Participants
  Low Risk | 1 | 2
  Medium Risk | 0 | 0
  High Risk | 0 | 0

45. Other Pre Specified Outcome: Columbia Suicide Severity Rating Scale (CSSRS)
Description: as for outcome 41
Time Frame: week 4 for patients age 17 or older
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1 | 1
Participants
  Low Risk | 0 | 1
  Medium Risk | 1 | 0
  High Risk | 0 | 0

46. Other Pre Specified Outcome: Columbia Suicide Severity Rating Scale (CSSRS)
Description: as for outcome 41
Time Frame: week 5 for patients age 17 or older
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1 | 1
Participants
  Low Risk | 0 | 1
  Medium Risk | 1 | 0
  High Risk | 0 | 0

47. Other Pre Specified Outcome: Columbia Suicide Severity Rating Scale (CSSRS)
Description: as for outcome 41
Time Frame: week 6 for patients age 17 or older
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1 | 0
Participants
  Low Risk | 0 | 0
  Medium Risk | 1 | 0
  High Risk | 0 | 0

48. Other Pre Specified Outcome: Columbia Suicide Severity Rating Scale (CSSRS)
Description: as for outcome 41
Time Frame: week 7 for patients age 17 or older
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

49. Other Pre Specified Outcome: Columbia Suicide Severity Rating Scale (CSSRS)
Description: as for outcome 41
Time Frame: week 8 for patients age 17 or older
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

50. Other Pre Specified Outcome: Columbia Suicide Severity Rating Scale (CSSRS)
Description: as for outcome 41
Time Frame: week 9 for patients age 17 or older
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

51. Other Pre Specified Outcome: Columbia Suicide Severity Rating Scale (CSSRS)
Description: as for outcome 41
Time Frame: 6 months after enrollment for patients age 17 or older
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

52. Other Pre Specified Outcome: Ask Suicide Screening Questions (ASQ)
Description: Evidence-based metric evaluating for presence of suicidal ideation and severity. Scores include 1 (negative screen), 2 (non-acute positive screen), and 3 (acute positive screen). Higher scores represent higher suicidal ideation and higher risk of suicide.
Time Frame: Measured at enrollment for patients age 16 or younger
Population: Numbers represent participants enrolled at this time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 2
Participants
  Negative Screen | 1 | 2
  Non-Acute Positive Screen | 3 | 0
  Acute Positive Screen | 0 | 0

53. Other Pre Specified Outcome: Ask Suicide Screening Questions (ASQ)
Description: as for outcome 52
Time Frame: week 1 for patients age 16 or younger
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 2
Participants
  Negative Screen | 1 | 1
  Non-Acute Positive Screen | 3 | 1
  Acute Positive Screen | 0 | 0

54. Other Pre Specified Outcome: Ask Suicide Screening Questions (ASQ)
Description: as for outcome 52
Time Frame: week 2 for patients age 16 or younger
Population: Numbers represent participants enrolled at this time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 2
Participants
  Negative Screen | 1 | 1
  Non-Acute Positive Screen | 3 | 1
  Acute Positive Screen | 0 | 0

55. Other Pre Specified Outcome: Ask Suicide Screening Questions (ASQ)
Description: as for outcome 52
Time Frame: week 3 for patients age 16 or younger
Population: Numbers represent participants enrolled at this time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 2
Participants
  Negative Screen | 1 | 1
  Non-Acute Positive Screen | 3 | 1
  Acute Positive Screen | 0 | 0

56. Other Pre Specified Outcome: Ask Suicide Screening Questions (ASQ)
Description: as for outcome 52
Time Frame: week 4 for patients age 16 or younger
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 2 | 2
Participants
  Negative Screen | 2 | 2
  Non-Acute Positive Screen | 0 | 0
  Acute Positive Screen | 0 | 0

57. Other Pre Specified Outcome: Ask Suicide Screening Questions (ASQ)
Description: as for outcome 52
Time Frame: week 5 for patients age 16 or younger
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 2 | 2
Participants
  Negative Screen | 1 | 2
  Non-Acute Positive Screen | 1 | 0
  Acute Positive Screen | 0 | 0

58. Other Pre Specified Outcome: Ask Suicide Screening Questions (ASQ)
Description: as for outcome 52
Time Frame: week 6 for patients age 16 or younger
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 2
Participants
  Negative Screen | 2 | 2
  Non-Acute Positive Screen | 1 | 0
  Acute Positive Screen | 0 | 0

59. Other Pre Specified Outcome: Ask Suicide Screening Questions (ASQ)
Description: as for outcome 52
Time Frame: week 7 for patients age 16 or younger
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

60. Other Pre Specified Outcome: Ask Suicide Screening Questions (ASQ)
Description: as for outcome 52
Time Frame: week 8 for patients age 16 or younger
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 1
Participants
  Low Risk | 2 | 1
  Medium Risk | 1 | 0
  High Risk | 0 | 0

61. Other Pre Specified Outcome: Ask Suicide Screening Questions (ASQ)
Description: as for outcome 52
Time Frame: week 9 for patients age 16 or younger
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 1
Participants
  Negative Screen | 2 | 1
  Non-Acute Positive Screen | 1 | 0
  Acute Positive Screen | 0 | 0

62. Other Pre Specified Outcome: Ask Suicide Screening Questions (ASQ)
Description: as for outcome 52
Time Frame: 6 months after enrollment for patients age 16 or younger
Population: Numbers represent participants enrolled at this time point, other participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 2 | 1
Participants
  Negative Screen | 2 | 1
  Non-Acute Positive Screen | 0 | 0
  Acute Positive Screen | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 33 weeks for each participant.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/4
Other Adverse Events (participants affected / at risk) | 3/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=5) | Control (N=4)
Motor Vehicle Accident (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Participant had a bone fracture in a car accident
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=5) | Control (N=4)
Increase in Medication (Psychiatric disorders) | 1 (1) | 0 (0) — Increase in antidepressant medication
Less Headaches (General disorders) | 1 (1) | 0 (0) — Participant experienced less headaches
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) — Participants experienced nausea
Headache (General disorders) | 0 (0) | 1 (1) — Participant experienced headache
Sweating (Endocrine disorders) | 1 (1) | 0 (0) — Participant experienced sweating
Sore throat, runny nose, congestion (Infections and infestations) | 0 (0) | 2 (2) — Participants experienced common cold-like symptoms: sore throat, runny nose, and congestion.
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1) — Participant experienced a urinary tract infection
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Participant experienced constipation
Fever (Immune system disorders) | 0 (0) | 1 (1) — Participant experienced a fever

LIMITATIONS AND CAVEATS:
Limitations and caveats include low participant sample and participant attrition. No outcome data collected for outcome measures 48, 49, 50, 51, and 59 because participants were lost to follow-up at those time points.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT05073679/Prot_SAP_003.pdf
  • Informed Consent Form (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT05073679/ICF_002.pdf